CLINICAL TRIAL: NCT03939780
Title: Comparison of [18F]RO-948, [18F]MK-6240, and [18F]AV-1451 TAU Radiopharmaceuticals in Patients With Alzheimer's Disease and Older Controls
Brief Title: Tau Tracer Comparison in Healthy Controls and Alzheimer's Disease Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moving to another institution with NIH grant relinquished.
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00193649; 1R21AG062314-01 (NIH)
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Healthy; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- Cohort 1 (Experimental): Subjects will be scanned twice (once with each of the tracers [18F]RO-948 and [18F]MK-6240)
  Interventions: Diagnostic Test: [F18]RO-948; Diagnostic Test: [F18]MK-6240
- Cohort 2A (No Intervention): No PET scans will be done. Previous [18F]AV-1451 scans of selected aged matched older cognitively healthy controls (OC) subjects from the Baltimore Longitudinal Study of Aging (BLSA) study (IRB00047185) will be reanalyzed.
- Cohort 2B1 - AD [18F]RO-948 and [18F]AV-1451 (Experimental): Alzheimer's Disease (AD) subjects who show high binding to the choroid plexus by a visual analog scale (high, low, and none) will be studied. Subjects with AD will be scanned twice: once with [18F]RO-948 and a second scan with [18F]AV-1451 in randomized order and within one month of each other.
  Interventions: Diagnostic Test: [F18]RO-948; Diagnostic Test: [F18]AV1451
- Cohort 2B2 - AD [18F]MK-6240 and [18F]AV-1451 (Experimental): AD subjects who show high binding to the choroid plexus by a visual analog scale (high, low, and none) will be studied. Subjects with AD will be scanned twice: once with [18F]MK-6240 and a second scan with [18F]AV-1451 in randomized order and within one month of each other.
  Interventions: Diagnostic Test: [F18]MK-6240; Diagnostic Test: [F18]AV1451
- Cohort 2B3 - OC [18F]RO-948 and [18F]AV-1451 (Experimental): OC subjects who show high binding to the choroid plexus by a visual analog scale (high, low, and none) will be studied. Subjects with OC will be scanned twice: once with [18F]RO-948 and a second scan with [18F]AV-1451 in randomized order and within one month of each other.
  Interventions: Diagnostic Test: [F18]RO-948; Diagnostic Test: [F18]AV1451
- Cohort 2B4 - OC [18F]MK-6240 and [18F]AV-1451 (Experimental): OC subjects who show high binding to the choroid plexus by a visual analog scale (high, low, and none) will be studied. Subjects with OC will be scanned twice: once with [18F]MK-6240 and a second scan with [18F]AV-1451 in randomized order and within one month of each other.
  Interventions: Diagnostic Test: [F18]MK-6240; Diagnostic Test: [F18]AV1451

INTERVENTIONS:
Diagnostic Test: [F18]RO-948 — Single radiotracer IV injection with subsequent emission scan
  Arms: Cohort 1; Cohort 2B1 - AD [18F]RO-948 and [18F]AV-1451; Cohort 2B3 - OC [18F]RO-948 and [18F]AV-1451
Diagnostic Test: [F18]MK-6240 — Single radiotracer IV injection with subsequent emission scan
  Arms: Cohort 1; Cohort 2B2 - AD [18F]MK-6240 and [18F]AV-1451; Cohort 2B4 - OC [18F]MK-6240 and [18F]AV-1451
Diagnostic Test: [F18]AV1451 — Single radiotracer IV injection with subsequent emission scan
  Arms: Cohort 2B1 - AD [18F]RO-948 and [18F]AV-1451; Cohort 2B2 - AD [18F]MK-6240 and [18F]AV-1451; Cohort 2B3 - OC [18F]RO-948 and [18F]AV-1451; Cohort 2B4 - OC [18F]MK-6240 and [18F]AV-1451

SUMMARY:
The primary objective of this study is to identify a new radioligand for imaging of tauopathy in Alzheimer's disease through direct comparisons of two potential candidates, [18F]RO-948 (formerly known as [18F]6958948) and [18F]MK-6240, and demonstration of the candidates' absence of off-target binding.

DETAILED DESCRIPTION:
This is an open label study to compare two new generation TAU radioligands, [18F]RO-948 (formerly known as [18F]6958948) and [18F]MK-6240, for imaging of tauopathy and demonstrate the radioligands' absence of off-target binding in patients with Alzheimer's disease (AD) and older healthy controls (OC). The study will directly compare AD and OC with these two next-generation TAU radio ligands and compare each of these radio ligands with the current most widely used first generation radioligand, [18F]AV-1451.

Up to 24 (12 AD and 12 OC, matched for age and sex with AD subjects) male and female subjects aged 50-100 will be enrolled in the study. The study consists of three cohorts.

* Cohort 1: 10 AD subjects and 10 aged and sex matched older controls will be enrolled. Subjects will be scanned twice, with each of the tracers [18F]RO-948 and [18F]MK-6240.
* Cohort 2A: No positron emission tomography (PET) scans will be done. Previous [18F]AV-1451 scans of selected aged matched OC subjects from the Baltimore Longitudinal Study of Aging (BLSA) study (IRB00047185) will be reanalyzed.
* Cohort 2B: 2 AD and 2 OC subjects who show high binding to the choroid plexus by a visual analog scale (high, low, and none) will be studied. Subjects will scanned twice with either: [18F]RO-948 or [18F]MK-6240 and a 2nd scan with [18F]AV-1451 in randomized order and within one month of each other.

ELIGIBILITY:
Inclusion Criteria (All):

* Male and female subjects 50 to 100 years of age
* Female subjects must be either surgically sterile or post-menopausal for at least 1 year or,
* Women of child bearing potential must commit to use a barrier contraception method for the duration of the study in addition to either an intra uterine device or hormonal contraception started at least 1 month prior to the first dose of radiotracer and until follow-up.
* Male subjects and their partners of childbearing potential must agree to use an effective method of contraception and will not donate sperm during the study. Barrier method must include use of a spermicide.
* Subjects who sign an IRB approved informed consent prior to any study procedures. Subjects deemed incapable of informed consent must provide assent and informed consent provided by, a legally authorized representative.
* Subjects who in the opinion of the investigator based on medical history and physical exam can tolerate the PET scan procedures.
* If subjects are on any concomitant medication, the indication and dosage of these medicines should be stable for at least 4 weeks prior to study start with the expectation that no relevant changes in use or dose will occur throughout the trial.
* Body mass index BMI between 18 and 32 kg per m2, Body weight less than 300 pounds.
* Normal cognitive function, including a normal Mini-Mental State Exam (MMSE) (>28) score as judged by the investigator for Control Subjects.

Inclusion Criteria for Subjects with a Diagnosis of Probable Alzheimer's disease

* Capacity for consent will be determined using the Alzheimer's Association Guidelines, developed at Johns Hopkins and described in Alzheimer's Association Consensus Recommendation Research consent for cognitively impaired adults Guidelines for Institutional Review Boards and Investigators Alzheimer's Association 2004.
* Have a reliable study partner able to accompany the subject to all visits and answer questions about the subject.
* Have a diagnosis of probable AD, according to the National Institute of Neurological and Communicative Disorders and Stroke Alzheimer's Disease and Related Disorders Association criteria
* MMSE score of between 16 and 26, inclusive.
* In the opinion of the investigator based on medical history and physical examination, can safely tolerate tracer administration and the scanning procedures.
* A positive visual read as per local procedures for florbetapir or similar procedures for other amyloid tracers of an amyloid PET scan, or amyloid-beta and tau cerebrospinal fluid (CSF) levels, which in the opinion of the principal investigator is consistent with a diagnosis of AD.

Exclusion Criteria:

* History or presence of a neurological diagnosis other than AD that may influence the outcome or analysis of the scan results examples include but are not limited to stroke, traumatic brain injury, space occupying lesions, non-Alzheimer's tauopathies, and Parkinson's disease.
* Subjects with a medical history that includes known autosomal dominant AD mutations in amyloid precursor protein (APP) or presenilin (PS) 1, PS 2 or mutations in genes that cause other types of autosomal dominant familial dementia, e.g., microtubule-associated protein tau (MAPT)
* History or presence of any clinically relevant hematological, hepatic, respiratory, cardiovascular, renal, metabolic, endocrine, or central nervous system (CNS) disease or other medical conditions that are not well controlled, may put the subject at risk, could interfere with the objectives of the study, or make the subject unsuitable for participation in the study for any other reason in the opinion of the principal investigator.
* Clinically relevant pathological findings in physical examination, ECG, or laboratory values at the screening assessment that could interfere with the objectives of the study.
* Known history of clinically significant infectious disease including AIDS or serological indication of acute or chronic hepatitis B or C or HIV infection.
* Women of childbearing potential must not be pregnant, or nursing and serum human chorionic gonadotropin (HCG) must be negative at the time of Screening Visit, and urine HCG must be negative on all subsequent visits.
* Loss or donation of more than 450 mL blood in the 4 months before screening or donation of plasma within 14 days of screening.
* Current symptoms of allergy and or severe allergy to drugs in medical history.
* History of drug or alcohol abuse or positive result from urine screen for drugs of abuse AD subjects on prescribed narcotics medications will not be excluded if urine drug screen is positive for the documented narcotic drugs.
* Have received an investigational medication within the last 3 months or 5 elimination half-life, whichever is longer, prior to administration of the radiotracer.
* Has had or is planning to have exposure to ionizing radiation that in combination with the study related tracer administrations and scanning procedures would result in a cumulative exposure that exceeds recommended exposure limits.
* Contraindications of MRI
* History of, or suffers from, claustrophobia or feels that he or she will be unable to lie still on their back in the MRI or PET scanner.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Tracer kinetics as measured by distribution volume of radioligands | 3 years
  Distribution volume (Vt) of the two newer radioligands, RO-948 and MK-6240, in older cognitively-normal control subjects (OC) and in clinically diagnosed Alzheimer's Disease (AD) patients.
Tracer kinetics as measured by Standard Uptake Volume Ratio of radioligands | 3 years
  Standard Uptake Volume Ratio (SUVR) of the two newer radioligands, RO-948 and MK-6240, in the OC and AD patients.
Tracer kinetics as measured by distribution volume of radioligands in off-target binding regions | 3 years
  Distribution volume (Vt) of the two newer radioligands, RO-948 and MK-6240, in older cognitively-normal control subjects (OC) and in clinically diagnosed Alzheimer's Disease (AD) patients in the off-target binding regions (basal ganglia, thalamus and choroid plexus).
Tracer kinetics as measured by SUVR of radioligands in off-target binding regions | 3 years
  SUVR of the two newer radioligands, RO-948 and MK-6240, in older cognitively-normal control subjects (OC) and in clinically diagnosed Alzheimer's Disease (AD) patients in the off-target binding regions (basal ganglia, thalamus and choroid plexus).

SECONDARY OUTCOMES:
Tracer kinetics as measured by distribution volume of radioligands in participants with high binding of AV-1541 | 3 years
  Distribution volume (Vt) of the two newer radioligands, RO-948 and MK-6240, in participants with confirmed high-binding of AV-1541 in choroid plexus
Tracer kinetics as measured by SUVR of radioligands in participants with high binding of AV-1541 | 3 years
  SUVR of the two newer radioligands, RO-948 and MK-6240, in participants with confirmed high-binding of AV-1541 in choroid plexus
Tracer kinetics as measured by volume distribution of radioligands in the hippocampus | 3 years
  Distribution volume (Vt) of the two newer radioligands, RO-948 and MK-6240, in older cognitively-normal control subjects (OC) and in clinically diagnosed Alzheimer's Disease (AD) patients in the hippocampus.
Tracer kinetics as measured by SUVR of radioligands in the hippocampus | 3 years
  SUVR of the two newer radioligands, RO-948 and MK-6240, in older cognitively-normal control subjects (OC) and in clinically diagnosed Alzheimer's Disease (AD) patients in the hippocampus.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Wong, MD/PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- John Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No